CLINICAL TRIAL: NCT03038139
Title: Changes in Spinal Muscular Activation and Creaniovertebral Angle After Postural Correction Program for Forward Head Posture
Brief Title: Postural Correction Exercises for Forward Head Posture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB- pGS- 2016-03- 144
Record Dates: First submitted 2017-01-23; First posted 2017-01-31 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-10

CONDITIONS: Forward Head Posture
Keywords: forward head posture; postural correction; spinal muscles

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cervical exercises (Experimental): Group A= Cervical correction program The cervical exercise program consist of 3 strengthening exercises and 2 stretching exercises.
  Applying exercises 3 times per week.
  Interventions: Other: Cervical exercises
- Lumbosacral exercises (Experimental): Group B= Cervical + Lumbosacral correction program The cervical exercise program consist of 3 strengthening exercises and 2 stretching exercises.
  The lumbosacral exercise program consist of 2 strengthening exercises and 4 stretching exercises.
  Applying exercises 3 times per week.
  Interventions: Other: Lumosacral exercises

INTERVENTIONS:
Other: Cervical exercises — Cervical correction program consist of 3 strengthening and 2 stretching exercises for neck and scapula Lumbosacral correction program consist of strengthening and stretching exercises for lumbar and sacral regions
  Arms: Cervical exercises
Other: Lumosacral exercises — Cervical and Lumbosacral correction program Lumbosacral program consist of 2 strengthening and 4 stretching exercises
  Arms: Lumbosacral exercises

SUMMARY:
The purpose of this study is to investigate the changes of spinal muscle activation in cervical, thoracic and lumbar segments for subjects with forward head posture (FHP) after application of two correction programs; a conventional one including cervical and thoracic spine, and a second program involving lumbosacral segment.

ELIGIBILITY:
Inclusion Criteria:

* adults with craniovertebral angle less than 50◦

Exclusion Criteria:

* Participants will be excluded if they have
* congenital spinal deformity such as scoliosis
* spinal conditions such as cervical trauma, fracture, instability of cervical spine, inflammation, infection, or neurological deficit
* a history of surgery at cervical spine or shoulder
* pregnant woman

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11; Primary Completion 2018-02 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Changes of Craniovertebral angle | 4 weeks
  The craniovertebral angle will be measure before and after 4 weeks of applying an exercise program.

SECONDARY OUTCOMES:
Electromyography | 4 weeks
  The Electromyography will be measure before and after 4 weeks of applying an exercise program.
Neck Disability Index | 4 weeks
  The neck disability index will be measure before and after 4 weeks of applying an exercise program.

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Dammam University, Dammam, Eastern Province
  - Dammam University, Dammam

IPD SHARING:
Plan to Share IPD: Undecided
only coded data (descriptive)

REFERENCES:
- See also: The effect of forward head posture on muscle activity during neck protraction and retraction — http://by7nn3rg6h.search.serialssolutions.com/?ctx_ver=Z39.88-2004&ctx_enc=info%3Aofi%2Fenc%3AUTF-8&rfr_id=info%3Asid%2Fsummon.serialssolutions.com&rft_val_fmt=info%3Aofi%2Ffmt%3Akev%3Amtx%3Ajournal&rft.genre=article&rft.atitle=The+effect+of+forward+head+posture+on+muscle+activity+during+neck+protraction+and+retraction&rft.jtitle=Journal+of+Physical+Therapy+Science&rft.au=Lee%2C+Kyeong-Jin&rft.au=Han%2C+Hee-Young&rft.au=Cheon%2C+Song-Hee&rft.au=Park%2C+So-Hyun&rft.date=2015&rft.issn=0915-5287&rft.eissn=2187-5626&rft.volume=27&rft.issue=3&rft.spage=977&rft.epage=979&rft_id=info:doi/10.1589%2Fjpts.27.977&rft.externalDBID=n%2Fa&rft.externalDocID=10_1589_jpts_27_977&paramdict=en-US
- See also: Changes in the activity of the muscles surrounding the neck according to the angles of movement of the neck in adults in their 20s — http://by7nn3rg6h.search.serialssolutions.com/?ctx_ver=Z39.88-2004&ctx_enc=info%3Aofi%2Fenc%3AUTF-8&rfr_id=info%3Asid%2Fsummon.serialssolutions.com&rft_val_fmt=info%3Aofi%2Ffmt%3Akev%3Amtx%3Ajournal&rft.genre=article&rft.atitle=Changes+in+the+activity+of+the+muscles+surrounding+the+neck+according+to+the+angles+of+movement+of+the+neck+in+adults+in+their+20s&rft.jtitle=Journal+of+Physical+Therapy+Science&rft.au=Lee%2C+Tae-Ho&rft.au=Lee%2C+Joon-Hyuk&rft.au=Lee%2C+Yun-Seob&rft.au=Kim%2C+Myoung-Kwon&rft.date=2015&rft.issn=0915-5287&rft.eissn=2187-5626&rft.volume=27&rft.issue=3&rft.spage=973&rft.epage=975&rft_id=info:doi/10.1589%2Fjpts.27.973&rft.externalDBID=n%2Fa&rft.externalDocID=10_1589_jpts_27_973&paramdict=en-US
- See also: Effect of an exercise program for posture correction on musculoskeletal pain — http://by7nn3rg6h.search.serialssolutions.com/?ctx_ver=Z39.88-2004&ctx_enc=info%3Aofi%2Fenc%3AUTF-8&rfr_id=info%3Asid%2Fsummon.serialssolutions.com&rft_val_fmt=info%3Aofi%2Ffmt%3Akev%3Amtx%3Ajournal&rft.genre=article&rft.atitle=Effect+of+an+exercise+program+for+posture+correction+on+musculoskeletal+pain&rft.jtitle=Journal+of+Physical+Therapy+Science&rft.au=Kim%2C+DeokJu&rft.au=Cho%2C+MiLim&rft.au=Park%2C+YunHee&rft.au=Yang%2C+YeongAe&rft.date=2015&rft.issn=0915-5287&rft.eissn=2187-5626&rft.volume=27&rft.issue=6&rft.spage=1791&rft.epage=1794&rft_id=info:doi/10.1589%2Fjpts.27.1791&rft.externalDBID=n%2Fa&rft.externalDocID=10_1589_jpts_27_1791&paramdict=en-US